CLINICAL TRIAL: NCT05498337
Title: Clinical Evaluation of Different Treatment Modalities for Vital Pulp of Immature Permanent Molars
Brief Title: Vital Pulp Therapy With Different Materials for Young Permanent Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nada mohamed, Assistant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vital pulp therapy
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Vital Pulp Therapy
Keywords: Alpexogenesis; MTA; Calcium hydroxide; Diode Laser
MeSH Terms: interventions — Calcium Hydroxide; Pemetrexed; Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Examiner (Other): Examiner
  Interventions: Other: calcium hydroxide; Other: MTA; Device: Diode Laser
- Patient (No Intervention): Patient

INTERVENTIONS:
Other: calcium hydroxide — Dental pulp medicament material
  Arms: Examiner
Other: MTA — Dental pulp medicament material
  Arms: Examiner
Device: Diode Laser — Device used in pulp therapy
  Arms: Examiner

SUMMARY:
This study will be conducted to:

Evaluate clinically and radiographically apexogenesis in immature permanent molars using:

1. Calcium Hydroxide.
2. MTA.
3. Laser.
4. Laser combined with MTA.

DETAILED DESCRIPTION:
Calcium Hydroxide has been the most commonly utilized pulpotomy agent for vital pulp therapy. It is the earliest medicament employed in pulpotomy that possesses the ability to stimulate tertiary dentinogenesis. This is attributed to its high alkalinity after mixing with water. Calcium hydroxide has a high pH, and its dental use relates chiefly to its ability to stimulate mineralization and also to its antibacterial property.

Biocompatibility and sealing ability are the most important properties, which account for optimal healing response in vital pulp therapy. Unlike conventional materials, MTA has low solubility and maintains its physical integrity after placement. It has several desirable characteristics in terms of biocompatibility, bioactivity, hydrophilicity, radiopacity, sealing ability and low solubility.

Diode laser in a young permanent tooth with traumatically exposed pulp has proved to be an effective technique for Pulpotomy in an immature tooth. Therefore, the use of soft-tissue diode lasers can influence the treatment outcome and should be seen as a predicable tool for vital pulp therapy.

ELIGIBILITY:
Inclusion Criteria:

* Medically free
* Vital teeth

Exclusion Criteria:

* Medically compromised
* Chronic abscess
* Non-vital teeth

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Root completion | one year
  Closure of radiographic apex using Scanora 5.2.6 digital software

SECONDARY OUTCOMES:
Root lengthening and thickening | one year
  Measuring the increase in length and width of the root canals using Scanora 5.2.6 digital software

OTHER OUTCOMES:
Clinical evaluation | one year
  Absence of pain and tenderness to percussion using facial scale

CONTACTS AND LOCATIONS:
Overall Officials: Salwa M Awad, Professor, Study Director — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakhalia Governrate, Egypt

IPD SHARING:
Plan to Share IPD: No